CLINICAL TRIAL: NCT03638349
Title: Actions & Insights Evaluating a Novel Diabetes Management Solution.
Acronym: ASCEND
Status: Completed | Type: Observational
Sponsor: LifeScan Scotland Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 3172697
Record Dates: First submitted 2018-07-26; First posted 2018-08-20 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus ( Type 1 and Type 2)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Single visit outcome study to obtain qualitative and quantitative data for a new BGMS.

DETAILED DESCRIPTION:
During ASCEND, patients will complete a single visit clinical study divided into two distinct parts. Part 1 involves each subject completing a number of simple quantitative exercises to gauge their level of comprehension of diabetes related information. Subjects will then continue during the same visit to complete part 2 which involves gathering qualitative feedback from each subject on the new Blood glucose monitoring system.

ELIGIBILITY:
Summary off:

Inclusion Criteria:

* Diagnosed with T1DM or T2DM
* Performs SMBG
* Male or female, at least 16 years old.
* Able to communicate (speak, read and write) in English
* Willing to sign an informed consent.

Exclusion Criteria:

* Unlikely to be compliant with the study in the opinion of study staff.
* Conflict of Interest - Prospective Participants are currently working for, previously worked for, or have an immediate family member currently working for a company that manufactures or markets the products tested under this procedure

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 150 male or female subjects with Type 1 or Type 2 Diabetes Mellitus.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Scaled preference questionnaires on new blood glucose monitoring digital tool. | 1 hour
  Proportion of positive responses from scaled response questionnaires, scaled from 1 to 6, 1 being the most negative response and 6 being the most positive.

SECONDARY OUTCOMES:
Scaled preference questionnaires on new blood glucose monitoring digital tool for Type 1 subjects. | 1 hour
  Proportion of positive responses from scaled response questionnaires, scaled from 1 to 6, 1 being the most negative response and 6 being the most positive.
Scaled preference questionnaires on new blood glucose monitoring digital tool for Type 2 subjects. | 1 hour
  Proportion of positive responses from scaled response questionnaires, scaled from 1 to 6, 1 being the most negative response and 6 being the most positive.
Scaled preference questionnaires on new blood glucose monitoring digital tool based on subject A1c. | 1 hour
  Proportion of positive responses from scaled response questionnaires, scaled from 1 to 6, 1 being the most negative response and 6 being the most positive.
Scaled preference questionnaires on new blood glucose monitoring digital tool based on subject subject numeracy. | 1 hour
  Proportion of positive responses from scaled response questionnaires, scaled from 1 to 6, 1 being the most negative response and 6 being the most positive.
Preference questionnaires on new blood glucose monitoring digital tool based on insulin or non-insulin using subjects | 1 hour
  Proportion of positive responses from scaled response questionnaires, scaled from 1 to 6, 1 being the most negative response and 6 being the most positive.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Grady, Study Director — LifeScan Scotland Ltd
Locations (3):
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Infirmary of Edinburgh, Edinburgh
  - Highland Clinical Research Facility, Inverness

IPD SHARING:
Plan to Share IPD: No